CLINICAL TRIAL: NCT01871818
Title: A Multi-centre Randomised Controlled Trial to Compare the Effectiveness of Two Rehabilitation Programs in Patients With Multiple Sclerosis.
Brief Title: A Trial to Compare the Effectiveness of Two Rehabilitation Programs for Multiple Sclerosis Patients
Acronym: REHABMUSCLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P110116
Record Dates: First submitted 2013-05-24; First posted 2013-06-07 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2017-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Rehabilitation; Chronic evolutive disease; Physiotherapy; Resistance training; Endurance training
MeSH Terms: conditions — Multiple Sclerosis | interventions — Physical Therapy Modalities; Private Practice

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combined program (Experimental): Combined program with physiotherapy, endurance training and resistance training.
  120 patients will receive this combined program
  Interventions: Behavioral: Combined program
- Physiotherapy (Active Comparator): Active comparator: physiotherapy in private practice 120 patients will receive this usual rehabilitation
  Interventions: Behavioral: Physiotherapy in private practice

INTERVENTIONS:
Behavioral: Combined program — Combined program with physiotherapy, endurance training and resistance training
  Arms: Combined program
Behavioral: Physiotherapy in private practice — Physiotherapy in private practice
  Arms: Physiotherapy

SUMMARY:
The purpose of this study was to compare the effectiveness of two rehabilitation programs (one month) in patients with multiple sclerosis. The first program is combined with physiotherapy, endurance training and resistance training. The second one is physiotherapy in private practice. Another purpose is to assess the length of the benefits of the combined program.

DETAILED DESCRIPTION:
This study will include 240 patients with a diagnosis of Multiple Sclerosis and with an Expanded Disability Status Scale ≤ 5. Patients will be divided into 2 groups, according to a randomization design. At recruitment (J0), after rehabilitation (M1) and at follow up (M3 and M6) each patient will be tested for the primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 year or over
* Able to walk independently without use of assistance 200 meters Expanded Disability Status Scale ≤5
* No relapse within the last three months
* No current or recent (six months) participation in intensive rehabilitation
* No recent modification (six months) of medications for MS
* Patients who received and signed information and informed consent

Exclusion Criteria:

* Cognitive impairments which could interfere with the ability to fully engage the rehabilitation program.
* Recent involvement (three months) in another interventional research study
* A complicating medical condition or orthopedic diagnosis that limits rehabilitation
* Cardiac or respiratory disease that interfere with endurance training
* Patient with safety measure
* Pregnant women, breastfeeding
* No affiliation to a social security

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2013-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test | 6 Minutes
  6 Minute Walk Test (6MWT) at the end of the rehabilitation program (Time Frame : at one month M1)

SECONDARY OUTCOMES:
Functional tests | 20 Minutes
  Functional tests: 10 meters Walk Test, Timed up and go test, Time to ascend and descend stairs, 6 Minute Walk Test
  Time frame:10 meters walk test = 2 min ; time up and going test= 4 min ; Time to ascend and descend stairs = 4 min ; et 6min walk = 6min
Aerobic capacity | 1h
  Aerobic capacity (V02 max)
Strength and fatigue of the knee flexors and extensors | 45 min
  Assessment of maximal voluntary strength using an isokinetic dynamometer or assessment of maximal voluntary strength using the 1-RM estimation
Clinical assessment | 45 min
  Spasticity assessment (Modified Ashworth Scale), passive range of motion of lower limb joint, lower limb strength (Medical Research Council scale), self questionnaire of pain.
Balance (Berg Balance scale) and postural control assessment | 15 min
Quality of Life assessment | 55 min
  Quality of Life assessed by self-reported questionnaire (SEP -59; EQ-5D), mood (HAD), MSIS-29, auto-questionnaire estimating the fatigue (Fatigue Severity Scale, Modified Fatigue Impact Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Djamel Bensmail, MD, Principal Investigator — Physical medicine and rehabilation Department, Hôpital RAYMOND POINCARE, 92380 Garches, France
Locations (1):
- Physical medicine and rehabilation Department, Hôpital RAYMOND POINCARE, Garches, Hauts DE Seine, France

REFERENCES:
- [Derived] Bonnyaud C, Hameau S, Zory R, Sznajder M, Heinzlef O, Aymard C, Chenet A, Medee B, Jacota M, Gallien P, Bensmail D; Rehabmuscle Team. Intensive interdisciplinary specialized rehabilitation or regular physiotherapy for multiple sclerosis? A randomised controlled trial with economic evaluation. Ann Phys Rehabil Med. 2025 Mar;68(2):101898. doi: 10.1016/j.rehab.2024.101898. Epub 2025 Jan 15. PMID 39818009